CLINICAL TRIAL: NCT05312866
Title: Intraoperative Retrolaminar Block as Opioid Free Anesthesia and Enhanced Recovery After Posterior Lumber Spine Discectomy: A Randomized Controlled Study
Brief Title: Intraoperative Retrolaminar Block as Opioid Free Anesthesia After Posterior Lumber Spine Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9325
Record Dates: First submitted 2022-03-27; First posted 2022-04-06 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Opioid Free Anesthesia
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard analgesia (paracetamol +fentanyl) (Active Comparator): Patients will receive standard analgesia (paracetamol 15mg/kg plus fentanyl 1ug/kg) iv
  Interventions: Procedure: Standard analgesia (paracetamol +fentanyl)
- Retrolaminar block with bupivacaine + magnesium sulfate + dexamethasone (Active Comparator): Patients will receive intraopertative retrolaminar block: 15 ml of bupivacaine 0. 25 % plus 2ml magnesium sulfate 10% (200mg) plus 2ml (8mg) dexamethasone on each side by slipping the needle of injection on the bone of spinous process and lamina.
  Interventions: Procedure: Retrolaminar block with bupivacaine + magnesium sulfate + dexamethasone

INTERVENTIONS:
Procedure: Standard analgesia (paracetamol +fentanyl) — Patients will receive standard analgesia (paracetamol 15mg/kg plus fentanyl 1ug/kg) iv
  Arms: Standard analgesia (paracetamol +fentanyl)
Procedure: Retrolaminar block with bupivacaine + magnesium sulfate + dexamethasone — Patients will receive intraopertative retrolaminar block: 15 ml of bupivacaine 0. 25 % plus 2ml magnesium sulfate 10% (200mg) plus 2ml (8mg) dexamethasone on each side by slipping the needle of injection on the bone of spinous process and lamina.
  Arms: Retrolaminar block with bupivacaine + magnesium sulfate + dexamethasone

SUMMARY:
Opioid-free intraoperative protocols have been successfully used in specific surgical populations with equal or superior results to classic general anesthetic approaches. In instances where opioid-free anesthesia may not be entirely feasible, there exists a continually growing body of evidence that the modern anesthesiologist has a potent pharmacologic and regional anesthetic arsenal that can reduce the amount of opioids required to effectively treat pain.

Retrolaminar block is considered a new, easy and simple technique with decreasing incidence of complications such as hypotension, pleural and nerve injury. Its efficacy had been investigated in trauma patients

DETAILED DESCRIPTION:
* Null hypothesis: Intraoperative retrolaminar block will not produce opioid sparing anesthetic effect and enhanced recovery after posterior lumber spine discectomy.
* Alternative hypothesis: Intraoperative retrolaminar block will produce opioid sparing anesthetic effect and enhanced recovery after posterior lumber spine discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Age: 21-60 years old.
* Sex: both sex (males and females).
* American Society of Anesthesiologist Physical status: ASA 1& II.
* Body Mass Index (BMI) = (25-30 kg/m2).
* Type of operation: elective posterior Lumbar discectomy from L3 to L5 disc space.

Exclusion Criteria:

* Altered mental state.
* Patients with known history of allergy to study drugs.
* Advanced hepatic, renal, cardiovascular, and respiratory diseases.
* Patients with chronic pain.
* Patients receiving anticoagulants.
* Contraindications of regional anesthesia, e.g., allergy to local anesthetics, coagulopathy, or septic focus at site of injection.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The recovery time | up to 1 hour postoperative
  The recovery time (time from discontinuation of isoflurane to first response to verbal command) will be recorded, then the patient will be transferred to the post anesthesia care unite (PACU) on standard monitors.

SECONDARY OUTCOMES:
pain intensity | up to 24 hours postoperative
  pain intensity measured using visual analogue scale from 0= no pain to 10= worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Human Medicine, Zagazig University, Zagazig, Alsharquia, Egypt